CLINICAL TRIAL: NCT00462397
Title: Phase II Study of Weekly Neoadjuvant Chemotherapy Followed by Radical Chemoradiation for Locally Advanced Cervical Cancer
Brief Title: Paclitaxel and Carboplatin Followed by Cisplatin and Radiation Therapy in Treating Patients With Stage IB, Stage II, Stage III, or Stage IVA Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College London Hospitals (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000540233; UCLCTC-BRD/05/22-CERVIX; EUDRACT-2005-000134-20; CRUK-BRD/05/22; EU-20720; UCLCTC-CERVIX
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2007-04

CONDITIONS: Cervical Cancer
Keywords: cervical adenocarcinoma; cervical adenosquamous cell carcinoma; cervical squamous cell carcinoma; stage IB cervical cancer; stage IIA cervical cancer; stage IIB cervical cancer; stage III cervical cancer; stage IVA cervical cancer; recurrent cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Carboplatin; Cisplatin; Paclitaxel; Neoadjuvant Therapy; Brachytherapy; Radiotherapy

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin
Drug: paclitaxel
Procedure: neoadjuvant therapy
Radiation: brachytherapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as paclitaxel, carboplatin, and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving combination chemotherapy together with radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving paclitaxel together with carboplatin followed by cisplatin and radiation therapy works in treating patients with stage IB, stage II, stage III, or stage IVA cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate, in terms of clinical or radiologic response at 12 weeks after completion of study therapy, in patients with stage IB2-IVA cervical cancer treated with neoadjuvant chemotherapy comprising dose-dense paclitaxel and carboplatin followed by radical chemoradiotherapy comprising concurrent cisplatin and radiotherapy.

Secondary

* Determine the response rate in patients treated with this neoadjuvant chemotherapy regimen.
* Determine the toxicity of this neoadjuvant chemotherapy regimen in these patients.
* Assess the progression-free survival of patients treated with this regimen.
* Determine the overall survival of patients treated with this regimen.

OUTLINE: This is a multicenter study.

* Neoadjuvant chemotherapy: Patients receive neoadjuvant chemotherapy comprising paclitaxel IV over 1 hour and carboplatin IV over 30 minutes on day 1. Treatment repeats weekly for up to 6 courses in the absence of disease progression or unacceptable toxicity.
* Chemoradiotherapy: Beginning in week 7, or as soon as blood counts recover, patients receive cisplatin IV over 1 hour on day 1. Treatment repeats weekly for 4-6 courses in the absence of disease progression or unacceptable toxicity. Patients also undergo concurrent radiotherapy comprising pelvic external beam radiotherapy once daily for 5½ weeks (5 weeks for patients with positive para-aortic lymph nodes) and 2 applications of high-dose rate intracavitary brachytherapy or low- or medium-dose rate brachytherapy. Patients with parametrial or pelvic sidewall disease extension also undergo external boost radiotherapy for 3 days.

After completion of study therapy, patients are followed periodically for 2 years.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed carcinoma of the cervix, including any of the following subtypes:

  * Squamous cell carcinoma
  * Adenocarcinoma
  * Adenosquamous cell carcinoma
* Locally advanced disease (i.e., FIGO stage IB2-IVA disease)

  * Stage confirmed by examination under anesthesia, cystoscopy, and sigmoidoscopy with biopsy of any suspicious lesions in the bladder, vagina, or rectum
* Disease suitable for treatment with radical intent using chemoradiotherapy

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Platelet count > 100,000/mm^3
* Hemoglobin > 12.5 g/dL
* WBC > 3,000/mm^3
* Absolute neutrophil count > 1,500/mm^3
* Bilirubin < 1.25 times upper limit of normal (ULN)
* Glomerular filtration rate (GFR) normal by ethylenediaminetetraacetic acid (EDTA) OR creatinine clearance ≥ 60 mL/min
* Placement of ureteric stents required for all patients with hydronephrosis, regardless of renal function
* ALT or AST < 2.5 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* No prior diagnosis of cancer, except basal cell skin cancer
* No active cardiac disease
* Deemed fit to receive chemoradiotherapy
* ECG normal

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-06

PRIMARY OUTCOMES:
Response rate at the end of chemoradiotherapy (i.e., 12 weeks after completion of study therapy)

SECONDARY OUTCOMES:
Response rate at the end of neoadjuvant treatment (i.e., 6 weeks after study entry)
Toxicity as assessed by NCI CTCAE v3.0
Progression-free survival
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Mary McCormack, MD, Study Chair — University College London Hospitals
Locations (3):
- United Kingdom (3):
  - Leicester Royal Infirmary, Leicester, England
  - Royal Marsden - London, London, England
  - University College of London Hospitals, London, England